CLINICAL TRIAL: NCT00163722
Title: A Multicentre Randomised Controlled Trial Comparing the Current Standard Diagnostic Strategy for Invasive Aspergillosis to the New Diagnostic Strategy for Invasive Aspergillosis in High-Risk Haematology Patients in Order to Determine Which Strategy Results in the Lower Rates of Use of Empiric Antifungal Therapy
Brief Title: A Multicentre Randomised Controlled Trial Comparing Two Strategies for the Diagnosis of Invasive Aspergillosis in High-risk Haematology Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 55/05; ALLG SC01; NHMRC Project Grant 331305
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2005-09

CONDITIONS: Invasive Aspergillosis
MeSH Terms: interventions — Culture Techniques; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard diagnostic strategy of culture and histology (Active Comparator): The standard-diagnostic strategy was designed to be consistent with the 2002 guidelines for antimicrobial use in neutropenic patients with cancer. When an invasive fungal infection was suspected (e.g. persistent fevers) cultures of blood, urine, sputum (if available) and faeces (if clinically indicated), and HRCT scans of chest were performed. Bronchoscopy and biopsies were performed according to institutional protocols. Empiric antifungal therapy was recommended whilst undergoing these investigations and was continued, de-escalated to prophylaxis, or changed to treatment of invasive aspergillosis or other IFD according to test results.
  Interventions: Other: Culture and histology
- Aspergillus galactomannan and PCR directed (Experimental): Results of once to twice weekly testing with Aspergillus galactomannan and PCR directed the timing of CT scan performance and whether antifungal therapy was given
  Interventions: Other: Aspergillus galactomannan and PCR

INTERVENTIONS:
Other: Culture and histology
  Arms: Standard diagnostic strategy of culture and histology
Other: Aspergillus galactomannan and PCR
  Arms: Aspergillus galactomannan and PCR directed

SUMMARY:
Aspergillus is a fungus found in soil, on farms and on construction sites. In those whose immune system is impaired it causes severe infection. The people who are particularly at high-risk of infection with Aspergillus (which is called Invasive Aspergillosis)are those with acute leukaemia who are having chemotherapy and those post bone marrow transplantation. Currently 15% of those at high-risk develop Invasive Aspergillosis and 60-90% of those with Invasive Aspergillosis die.

The main reason for this high death rate is that our current diagnostic tests are not good at detecting infection or often only detect the infection at advanced stages when treatment is ineffective. Because of the limitations of current diagnostic tests the current practice is to give empiric antifungal therapy (EAFT) early to treat suspected Invasive Aspergillosis. However studies have demonstrated that this therapy has only resulted in a minor reduction in the mortality rates and it also causes significant drug toxicity. It is a suboptimal treatment modality.

New tests have recently been developed to diagnose Invasive Aspergillosis. These tests are for the detection of an Aspergillus protein in blood and for the detection of Aspergillus DNA in blood. Available data suggests that these new tests make an early diagnosis and seem to be able to monitor responses to treatment. However no study has been reported to date which demonstrates that the use of these tests can impact on important patient outcomes. This trial is being performed to determine whether the use of the new diagnostic tests to guide antifungal therapy will help improve treatment of Invasive Aspergillosis, reduce drug toxicity and reduce the death rate in the high-risk patients as compared with the current standard method of diagnosis and treatment with EAFT.

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling all the following criteria will be eligible for enrolment 1. Aged 18-80 years 2. Undergoing allogeneic haematopoietic stem cell transplantation (HSCT) for any reason OR Undergoing intensive combination chemotherapy for acute myeloid leukaemia (AML) or acute lymphoblastic leukaemia (ALL) 3. Has given written informed consent.

-

Exclusion Criteria:

Patients with any of the following will be ineligible for enrolment 1. Other immunocompromised states (e.g. HIV infection, solid organ transplantation, autoimmune conditions treated with immunosuppressants etc.) besides those outlined in the inclusion criteria above 2. Currently enrolled in an antifungal treatment trial (not an antifungal prophylaxis trial) 3. Past history of proven or probable IA (as per standardized definitions) during a previous cycle of chemotherapy 4. Currently have active IA or other active invasive fungal infection 5. Prior enrolment in this study

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2005-09; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The proportion of patients treated with at least 1 course of empiric antifungal therapy as per protocol definition at 26 weeks following randomisation | 26 weeks of follow-up

SECONDARY OUTCOMES:
Invasive Aspergillosis related mortality rates | 26 weeks of follow-up
Other invasive fungal infection-related (IFI) mortality rates | 26 weeks of follow-up
All-cause mortality rates | 26 weeks of follow-up
Nephrotoxicity rates | 26 weeks of follow-up
Hepatotoxicity rates | 26 weeks of follow-up
Total number of courses of empiric antifungal therapy | 26 weeks of follow-up
Cost data associated with treatment and complications. | 26 weeks of follow-up
  To include number of hospital admissions, hospital length of stay, total duration of antifungal therapy and number of invasive procedures to diagnose invasive aspergillosis
Incidence of proven, probable and possible invasive aspergillosis | 26 weeks of follow-up
Incidence of proven, probable and possible other invasive fungal disease besides invasive aspergillosis | 26 weeks of follow-up

OTHER OUTCOMES:
Sub-group analysis according to type of antifungal prophylaxis, underlying disease and centre | 26 weeks of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Monica Slavin, MB BS FRACP, Principal Investigator — Infectious Diseases Unit, Peter MacCallum Cancer Centre, St. Andrew's Place, East Melbourne, Victoria, Australia; Orla Morrissey, MB BCh FRACP, Principal Investigator — Infectious Diseases Unit, Alfred Hospital, Level 2, Burnet Institute, Commercial Road, Melbourne, Victoria, 3004, Australia
Locations (6):
- Australia (6):
  - St. Vincent's Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria

REFERENCES:
- [Derived] Morrissey CO, Chen SC, Sorrell TC, Milliken S, Bardy PG, Bradstock KF, Szer J, Halliday CL, Gilroy NM, Moore J, Schwarer AP, Guy S, Bajel A, Tramontana AR, Spelman T, Slavin MA; Australasian Leukaemia Lymphoma Group and the Australia and New Zealand Mycology Interest Group. Galactomannan and PCR versus culture and histology for directing use of antifungal treatment for invasive aspergillosis in high-risk haematology patients: a randomised controlled trial. Lancet Infect Dis. 2013 Jun;13(6):519-28. doi: 10.1016/S1473-3099(13)70076-8. Epub 2013 Apr 30. PMID 23639612
- [Derived] Morrissey CO, Chen SC, Sorrell TC, Bradstock KF, Szer J, Halliday CL, Gilroy NM, Schwarer AP, Slavin MA. Design issues in a randomized controlled trial of a pre-emptive versus empiric antifungal strategy for invasive aspergillosis in patients with high-risk hematologic malignancies. Leuk Lymphoma. 2011 Feb;52(2):179-93. doi: 10.3109/10428194.2010.542600. PMID 21281234